CLINICAL TRIAL: NCT07384455
Title: Comparıson of the effectıveness of ephedrıne and norepınephrıne ın the Treatment of hypotensıon developıng ın spınal anaesthesıa durıng Caesarean sectıon surgerıes
Brief Title: Use of Vasopressors in Hypotension Associated With Spinal Anaesthesia in Caesarean Sections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, M.D, co-investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-24695
Record Dates: First submitted 2026-01-16; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Caesarean Section
Keywords: spinal anesthesia; Hypotension; Norepinephrine
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Prospective randomize study
Masking Description: Prospective randomize study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 mg ephedrine intravenously after spinal anaesthesia (Experimental): Group 1: Group administered 10 mg ephedrine intravenously after spinal anaesthesia
  Interventions: Procedure: Patients who received 10 mg of ephedrine intravenously after spinal anaesthesia during caesarean section
- 8 mcg of norepinephrine intravenously following spinal anaesthesia (Experimental): Group 2: The group administered 8 mcg of norepinephrine intravenously following spinal anaesthesia
  Interventions: Procedure: Patients who received 8 mcg intravenous norepinephrine after spinal anaesthesia during caesarean section

INTERVENTIONS:
Procedure: Patients who received 10 mg of ephedrine intravenously after spinal anaesthesia during caesarean section — To prevent intraoperative hypotension, researchers administered 10 mg intravenous ephedrine to a group of patients after spinal anaesthesia.
  Arms: 10 mg ephedrine intravenously after spinal anaesthesia
Procedure: Patients who received 8 mcg intravenous norepinephrine after spinal anaesthesia during caesarean section — To prevent intraoperative hypotension, researchers administered 8 mcg intravenous norepinephrine to a group of patients after spinal anaesthesia.
  Arms: 8 mcg of norepinephrine intravenously following spinal anaesthesia

SUMMARY:
This study was designed as a prospective randomised study. In this study, the researchers planned to evaluate the effect of intravenous vasopressor agents administered to patients undergoing caesarean section under spinal anaesthesia on the incidence of hypotension. Our other aim was to evaluate perioperative haemodynamic data, maternal side effects and neonatal outcomes.

DETAILED DESCRIPTION:
Caesarean section is a significant procedure in obstetric patients and constitutes the vast majority of such operations. Regional anaesthesia is currently used in these patients, predominantly spinal anaesthesia. Considering the maternal and foetal side effects of hypotension associated with spinal anaesthesia, it is necessary to prevent this. Vasopressors such as phenylephrine, ephedrine and norepinephrine are used for this purpose. To this end, the researchers aimed to evaluate the effect of ephedrine or norepinephrine administered in patients undergoing caesarean section under spinal anaesthesia on the incidence of hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients aged 18-45
* Pregnant patients with ASA 2
* Healthy pregnant women with a gestational age of 37-41 weeks

Exclusion Criteria:

* Pregnant patients with >ASA III Emergency cases multiple pregnancy preterm pregnancy pregnant women with foetal anomaly and placental anomaly those diagnosed with pre-eclampsia and eclampsia those with maternal cardiovascular and cerebrovascular disease body mass index > 40 kg/m² pregnant women with contraindications for spinal anaesthesia and who do not consent to the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
intraoperative hypotension | Intraoperative
  Our primary objective was to compare the incidence of intraoperative hypotension. In the study, hypotension was defined as a blood pressure level lower than 80% of the baseline systolic arterial pressure (SAP). Hypotension was determined in both groups when the systolic arterial pressure was lower than 80% despite the administration of ephedrine or norepinephrine after spinal anaesthesia
Assessment of intraoperative heart rate | intraoperative
  Our secondary objective is to assess the intraoperative heart rate. These time intervals were at the start of surgery, after the patient was placed in the sitting position, after spinal anaesthesia was administered, 3 minutes, 6 minutes, 9 minutes, 12 minutes, and 15 minutes after spinal anaesthesia, 1 minute after delivery, 10 minutes, 20 minutes, 30 minutes, and 40 minutes after delivery, and at the end of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Mushambi MC, Kinsella SM, Popat M, Swales H, Ramaswamy KK, Winton AL, Quinn AC; Obstetric Anaesthetists' Association; Difficult Airway Society. Obstetric Anaesthetists' Association and Difficult Airway Society guidelines for the management of difficult and failed tracheal intubation in obstetrics. Anaesthesia. 2015 Nov;70(11):1286-306. doi: 10.1111/anae.13260. PMID 26449292
- [Result] Singh PM, Singh NP, Reschke M, Ngan Kee WD, Palanisamy A, Monks DT. Vasopressor drugs for the prevention and treatment of hypotension during neuraxial anaesthesia for Caesarean delivery: a Bayesian network meta-analysis of fetal and maternal outcomes. Br J Anaesth. 2020 Mar;124(3):e95-e107. doi: 10.1016/j.bja.2019.09.045. Epub 2019 Dec 4. PMID 31810562
- [Result] Massoth C, Topel L, Wenk M. Hypotension after spinal anesthesia for cesarean section: how to approach the iatrogenic sympathectomy. Curr Opin Anaesthesiol. 2020 Jun;33(3):291-298. doi: 10.1097/ACO.0000000000000848. PMID 32371631
- [Result] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Result] Allen TK, George RB, White WD, Muir HA, Habib AS. A double-blind, placebo-controlled trial of four fixed rate infusion regimens of phenylephrine for hemodynamic support during spinal anesthesia for cesarean delivery. Anesth Analg. 2010 Nov;111(5):1221-9. doi: 10.1213/ANE.0b013e3181e1db21. Epub 2010 May 21. PMID 20495139
- [Result] Park HS, Choi WJ. Use of vasopressors to manage spinal anesthesia-induced hypotension during cesarean delivery. Anesth Pain Med (Seoul). 2024 Apr;19(2):85-93. doi: 10.17085/apm.24037. Epub 2024 Apr 30. PMID 38725163